CLINICAL TRIAL: NCT06613555
Title: Retinal Microvascularization in OCT-angiography and Systemic Diseases
Acronym: OCTAVA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ARNOULD 2022
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Systemic Vascular Damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with systemic vascular disease: * patients with either:
  * systemic vascular pathology
  * high cardiovascular risk
  * inflammatory vascular pathology
  * preeclampsia during pregnancy
  Interventions: Other: Retinal imaging; Biological: Biological check-up
- healthy controls: patients with no systemic or vascular inflammatory pathology and no high cardiovascular risk
  Interventions: Other: Retinal imaging; Biological: Biological check-up

INTERVENTIONS:
Other: Retinal imaging — the retinal imaging work-up includes:
  * OCT-angiography
  * Retinophotography
  * Adaptive optics
  performed at inclusion, at 6 months and then once a year for 10 years for patients Only performed at inclusion for controls
Biological: Biological check-up — it is performed at inclusion and then once a year for 10 years for patients
  Only performed at inclusion for controls

SUMMARY:
Systemic diseases are inflammatory, chronic illnesses affecting different organs and altering their function. At present, there are few non-invasive methods for predicting their onset and progression.

Some chronic diseases can be anticipated earlier thanks to predictive indicators. These indicators could help doctors decide which treatment is best suited to each patient. In particular, the state of microcirculation in the eyes, specifically in the retina, is linked to the progression of certain diseases in the body. Unfortunately, assessing the health of the small blood vessels in the retina is complicated. Most current methods are imprecise, difficult to reproduce and require qualified specialists. However, the use of retinal microcirculation appears to be a promising approach to solving these problems.

In fact, the structure of retinal blood vessels can be observed easily, painlessly and without invasive procedures, thanks to fundus photographs or scans providing imaging slices known as optical coherence tomography-angiography (OCT-A).

The vascularization of the retina is very often presented as a window giving access to the peripheral vascularization (the vascularization of other organs distant from the eyes).

For example, we recently demonstrated a link between retinal vascularization and the risk of heart problems in patients with coronary artery disease.

The aim of this study is to gather original information on the evolution of retinal vascularization, using specific markers that may be associated with damage to distant organs.

By regularly monitoring these changes over time, the researchers hope to identify early changes that could indicate the development or evolution of these diseases.

The main aim of this study is to create a database of images obtained by OCT-Angiography in patients with systemic diseases and in healthy individuals. This will enable us to identify early changes in retinal vascularization that may be associated with these systemic pathologies.

With this information, we hope to improve early diagnosis and monitoring of diseases, which could have a positive impact on patients' health.

ELIGIBILITY:
Inclusion Criteria:

For the "patients with systemic vascular disease" group

* Patients who have given oral, free and informed consent
* Patients with either :

  * systemic vascular pathology
  * high cardiovascular risk
  * inflammatory vascular pathology
  * preeclampsia during pregnancy

The study will also be offered to patients who have already had an OCT-A examination as part of their routine care, in order to follow them over time.

For the "healthy control" group

* Patients who have given free, oral and informed consent
* Patients with no prior systemic or vascular inflammatory pathology, and no high cardiovascular risk
* Non-diabetic patients
* Pregnant patients with risk-free pregnancies recruited from the gynecology department of CHU Dijon Bourgogne OR
* Adult patients without maculopathy recruited from the Ophthalmology Department of CHU Dijon Bourgogne

Exclusion Criteria:

* For the "patients with systemic vascular disease" group
* Ophthalmological history in both eyes (vascular and degenerative macular pathologies)
* Protected patient :

  * Minor patient
  * Patient under legal protection (guardianship, curatorship, court order)
  * Patient unable to give consent Person not affiliated to a social security scheme
  * Breast-feeding women
* Person with a contraindication to Tropicamide
* OCT-A signal strength < 7

For the "healthy control" group

* Any pathology studied in the case group
* Ophthalmological history in both eyes (vascular and degenerative macular pathologies)
* Type 1 or type 2 diabetes
* Person with a contraindication to Tropicamide
* Protected person :

  * Minor
  * Person under legal protection (guardianship, curatorship, court order)
  * Person unable to give consent
  * Person not affiliated to a social security scheme
  * Breast-feeding women
* OCT-A signal strength < 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic vascular disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2044-06 (Estimated); Study Completion 2044-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the evolution of retinal microvascular densities in OCT-A | Up to 10 years
Comparison of the clinical course of patients with systemic pathologies | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France